CLINICAL TRIAL: NCT00300313
Title: PTSD Prevention Using Escitalopram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Joseph Zohar, Prof. Joseph Zohar, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SHEBA-06-3913-JZ-CTIL
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Escitalopram
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — 10 to 20 mg / day
  Arms: 1
Drug: Placebo — 1-2 capsules
  Arms: 2

SUMMARY:
Assessing the efficacy of escitalopram in preventing the development of PTSD, or or reducing its severeness, after exposure to a traumatic event.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is able to read and understand the Patient Informed Consent.
2. The patient has signed the Patient Informed Consent.
3. The patient has sufficient knowledge of Hebrew in order to understand the study procedure and instruments
4. The patient is male or female aged between 18 and 65 years (extremes included).
5. The patient underwent a traumatic event, such as vehicle or other accident, terror attack, physical or sexual assault within the last 3 weeks, and no more than 4 weeks ago.
6. The patient meets either of the following criteria:

1. Full DSM-IV criteria for ASD 2. Intrusion and hyperarousal criteria only

Exclusion Criteria:

1. The patient refuses having any medication therapy. This patient will be referred to another treatment outside the study frame.
2. The patient has a serious physical injury at inclusion, in which his Abbreviated Injury Scale (AIS) score, for at least one of his body regions, is 3 or more, or that according to the judgment of the clinician his injury sequelae would interfere with the study treatment.
3. The patient uses concomitant medications not allowed in the study:

   1. Antidepressants, including MAOI, RIMA within the last 3 weeks prior to screening.
   2. Mood stabilizers within the last 3 weeks prior to screening.
   3. Antipsychotic medications within the last 3 weeks prior to screening.
   4. Anxiolytics 2 weeks in a row before randomization. Patient can participate in the study if did not take the medications for 3 days over the two weeks before randomization. Except for oxazepam 10-20 mg/day no more than 7 days in a raw.
   5. Serotonergic agonists (e.g. triptans) within the last 2 weeks prior to screening.
   6. Prophylactic treatment with any anticonvulsant drug.
   7. Herbal remedies that are psychoactive (e.g. St John's Wort, Kava kava, valerian, gingko biloba) within the last 3 weeks prior to screening.
4. The patient meets lifetime DSM-IV-TR criteria for:

   1. Mania or Bipolar disorder
   2. Schizophrenia
   3. Any personality disorder judged by the investigator to jeopardize the evaluation of the treatment.
   4. Mental retardation or pervasive disorder
   5. Cognitive disorder (inc. dementia)
5. The patient has or has had alcohol or drug abuse related disorders in the last year prior to the screening visit.
6. The patient has, in the investigator's opinion, significant suicide risk and/or a score of ≥ 5 on question 10 in the MADRS scale.
7. The patient has a history of severe suicide attempt.
8. The patient requires ElectroConvulsive Therapy (ECT) or has received ECT within the last year prior to the screening visit.
9. The patient is currently serving in the Israeli security forces.
10. The patient has a history of drug allergy or hypersensitivity, or known hypersensitivity to escitalopram or citalopram.
11. The patient has an illness and/or serious sequelae thereof, severe enough according to the clinician judgment, to prevent his participation in the study, including liver or renal insufficiency; cardiovascular, pulmonary, gastrointestinal, endocrine (inc. uncontrolled thyroid), neurological (inc. epilepsy), infectious, neoplastic, or metabolic disturbances
12. The patient is pregnant or breast-feeding.
13. The patient, if woman of childbearing potential, is not using adequate contraception (adequate contraception is defined as sexual abstinence, oral/systemic contraception, surgical sterilisation, intrauterine device, diaphragm in combination with spermicide, or condom for male partner in combination with spermicide).
14. The patient, in the opinion of the investigator, is unlikely to comply with the clinical study protocol.
15. The patient has previously participated in the current study or in any other study within the last 30 days.
16. The patient has familial relationships with the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
CAPS | 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Study Director — Chaim Sheba Medical Center
Locations (5):
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - RAMBAM Medical Center, Haifa
  - Hadassa Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan

REFERENCES:
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873
- [Derived] Zohar J, Fostick L, Juven-Wetzler A, Kaplan Z, Shalev H, Schreiber G, Miroshnik N, Shalev AY, Stein DJ, Seedat S, Suliman S, Klein E. Secondary Prevention of Chronic PTSD by Early and Short-Term Administration of Escitalopram: A Prospective Randomized, Placebo-Controlled, Double-Blind Trial. J Clin Psychiatry. 2018 Mar/Apr;79(2):16m10730. doi: 10.4088/JCP.16m10730. PMID 28703951
- [Derived] Suliman S, Seedat S, Pingo J, Sutherland T, Zohar J, Stein DJ. Escitalopram in the prevention of posttraumatic stress disorder: a pilot randomized controlled trial. BMC Psychiatry. 2015 Feb 19;15:24. doi: 10.1186/s12888-015-0391-3. PMID 25885650